CLINICAL TRIAL: NCT01910480
Title: A Phase 1, Open-Label Study to Assess the Effect of Ketoconazole on the Pharmacokinetics of NBI-98854 in Healthy Subjects
Brief Title: Study to Assess the Effect of Ketoconazole on the Pharmacokinetics of NBI-98854 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NBI-98854-1302
Record Dates: First submitted 2013-07-24; First posted 2013-07-29 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Effect of Ketoconazole on the PK of NBI-98854 in Healthy Subjects
MeSH Terms: interventions — valbenazine; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NBI-98854 followed by NBI-98854 with ketoconazole (Experimental): 50 mg NBI-98854 on Study Days 1 and 6 and 200 mg ketoconazole twice daily on Study Days 5 through 9.
  Interventions: Drug: NBI-98854 50 mg capsule once daily; Drug: Ketoconazole 400 mg (200 mg twice daily)

INTERVENTIONS:
Drug: NBI-98854 50 mg capsule once daily
Drug: Ketoconazole 400 mg (200 mg twice daily)

SUMMARY:
The purposes of this study are to: learn about the safety of the study drug (NBI-98854); learn how subjects tolerate the study drug; and evaluate and compare the pharmacokinetics (PK testing, the study of how the body absorbs, distributes, breaks down and eliminates a drug) of the investigational study drug after taking it alone and with ketoconazole. Ketoconazole is known to affect the PK of many drugs and is studied to more safely prescribe medications.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteer, 18 to 40 years of age.
* Subjects of childbearing potential must agree to use hormonal or two forms of nonhormonal birth control during the study.
* Female subjects must not be pregnant, given birth within 1 year of study start, or breastfeeding.
* Be in good general health and expected to complete the clinical study as designed.
* Have a body mass index (BMI) of 18 to 30 kg/m2 (both inclusive).

Exclusion Criteria:

* Have an active clinically significant unstable medical condition within 1 month (30 days) prior to screening.
* Have a history of substance dependence or substance (drug) or alcohol abuse within the 3 months before study start.
* Report more than two alcoholic beverages daily or more than 14 alcoholic beverages weekly withing 7 days of study start.
* Report use of tobacco and/or nicotine-containing products within 3 months of study start.
* Have a known history of neuroleptic malignant syndrome.
* Have a significant risk of suicidal or violent behavior.
* Have a positive human immunodeficiency virus antibody, (HIV-Ab), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody result at screening or have a history of positive result.
* Have received an investigational drug within 30 days before screening or plan to use an investigational drug (other than NBI-98854) during the study.
* Have an allergy, hypersensitivity, or intolerance to tetrabenazine.
* Had a blood loss greater than or equal to 500 mL or donated blood within 56 days of study start.
* Have had previous exposure with NBI-98854.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of plasma concentrations of NBI-98854 and metabolites following administration of NBI-98854 alone | 45 minutes prior to NBI-98854 dosing, and at 15, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 48, 72 and 96 hours postdose
Evaluation of plasma concentrations of NBI-98854 and metabolites following administration of NBI-98854 concomitantly with ketoconazole | at 45 minutes prior to NBI-98854 dosing, and at 15, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 48, 72 and 96 hours postdose
Number of Participants with Adverse Events following dosing with NBI-98854 | Up to 31 days

CONTACTS AND LOCATIONS:
Overall Officials: Chris O'Brien, MD, Study Director — Neurocrine Biosciences
Locations (1):
- Celerion, Tempe, Arizona, United States